CLINICAL TRIAL: NCT06859294
Title: A Phase 2a, Single-Arm Study to Investigate the Efficacy and Safety of LY3541860 in Adult Participants With Moderately to Severely Active Rheumatoid Arthritis
Brief Title: A Study of LY3541860 in Adult Participants With Moderately to Severely Active Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27372; J3K-MC-KIAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3541860 (Experimental): LY3541860 will be administered intravenously (IV).
  Interventions: Drug: LY3541860

INTERVENTIONS:
Drug: LY3541860 — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the effects of LY3541860 in adult participants with moderately to severely active Rheumatoid Arthritis with inadequate response to a least one biologic disease-modifying antirheumatic drug (bDMARD)or targeted synthetic disease-modifying antirheumatic drug (tsDMARD).

Study participation is approximately 50 weeks, including a 6-week screening period, 24-week treatment period, and a 20-week safety follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset Rheumatoid Arthritis (RA) for at least 3 months prior to screening, as defined by the 2010 ACR/EULAR classification criteria.
* Have moderately to severely active RA, at screening (Visit 1) and baseline (Visit 2), defined by the presence of

  * ≥6 swollen joints based on 66 joint count (and ≥4 swollen joints on 28 joint count), and
  * ≥6 tender joints based on 68 joint count (and ≥4 tender joints on 28 joint count).
* Have active synovitis in ≥1 joint, in hands or wrists, of the investigator choosing at screening, having an MRI synovitis RAMRIS score of ≥2 as determined from the central reading of the images.

Exclusion Criteria:

* Have a diagnosis or history of malignant disease within 5 years prior to baseline, with the exceptions of

  * basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years, or
  * cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to baseline.
* Have estimated glomerular filtration rate (eGFR) of <45 milliliter per minute (mL/minute) from serum creatinine using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation.
* Have a current or recent active infection.
* Have presence of 1 or more significant concurrent medical conditions per investigator judgment, including but not limited to

  * poorly controlled diabetes or hypertension
  * chronic kidney disease Stage 3a or b, 4, or 5
  * symptomatic heart failure according to New York Heart Association Class 2, 3, or 4
  * myocardial infarction, unstable angina pectoris, stroke, or transient ischemic attack within the past 12 months before baseline
  * severe chronic pulmonary disease, for example, requiring oxygen therapy major chronic inflammatory disease or connective tissue disease other than RA, including but not limited to
  * systemic lupus erythematosus
  * psoriatic arthritis
  * axial spondyloarthritis, including ankylosing spondylitis and non-radiographic axial spondyloarthritis
  * reactive arthritis
  * gout
  * scleroderma
  * polymyositis
  * dermatomyositis
  * active fibromyalgia, or
  * multiple sclerosis
* Have received any prior B-cell targeted therapy (for example, anti-CD19 antibodies or anti-CD20 antibodies, such as rituximab).
* Received corticosteroids, opioids, conventional disease-modifying antirheumatic drug (cDMARD), with changes in dose or have received Janus kinase (JAK) inhibitors within 28 days prior to the screening MRI or plan on receiving these drugs during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Disease Activity Score - High-Sensitivity C-Reactive Protein (DAS28 - hsCRP) | Baseline, Week 12
  DAS28-hsCRP measures disease activity in 28 joints using a composite numeric score. Total scores range from 1.0 to 9.4, where a lower score indicates less disease activity.

SECONDARY OUTCOMES:
Change from Baseline in Rheumatoid Arthritis Magnetic Resonance Imaging Score (RAMRIS) Synovitis Score | Baseline, Week 12
  RAMRIS synovitis score ranges from 0-24, where a lower score indicates a lower level of inflammation.
Percentage of Participants Achieving American College of Rheumatology (ACR) 20 | Week 12
  ACR20 Responder is a participant who has at least 20% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity using VAS, Patient's Global Assessment of Disease Activity using VAS, HAQ-DI, pain due to arthritis, and hsCRP.
Percentage of Participants Achieving American College of Rheumatology (ACR) 50 | Week 12
  ACR50 Responder is a participant who has at least 50% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, HAQ-DI, pain due to arthritis, and hsCRP.
Percentage of Participants Achieving American College of Rheumatology (ACR) 70 | Week 12
  ACR70 Responder is a participant who has at least 70% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, HAQ-DI, pain due to arthritis, and hsCRP.
Change from Baseline in Disease Activity Score - Erythrocyte Sedimentation Rate (DAS28 - ESR) | Baseline, Week 12
  DAS28-ESR measures disease activity in 28 joints using a composite numeric score. Total scores ranged from 1.0-9.4, where lower scores indicated less disease activity.
Percentage of Participants Achieving Low disease activity (LDA) or Remission in Disease Activity Score - high-sensitivity C-reactive protein (DAS28-hsCRP) | Week 12
  DAS28-hsCRP measures disease activity in 28 joints using a composite numeric score. Total scores range from 1.0 to 9.4, where a lower score indicates less disease activity. The DAS28-hsCRP LDA is defined as DAS28-hsCRP ≤3.2.
Percentage of Participants Achieving European League Against Rheumatism (EULAR) Good Response Criteria | Week 12
  EULAR Responder index based on 28 joint counts categorizes clinical response based on improvement since baseline in DAS28-hsCRP. DAS28-CRP scores range from 1.0-9.4, where lower scores indicated less disease activity. EULAR DAS28-hsCRP responder index defines good response criteria as change in DAS28-hSCRP > 1.2 from baseline with a new DAS28 score <=3.2.
Change from Baseline in ACR Core Set Values Patient's Assessment of Arthritis Pain Using Visual Analog Scale (VAS) | Baseline, Week 12
  Participants were asked to assess their current level of arthritis pain by marking a vertical tick on a 100-mm horizontal VAS with the left end (0 mm) marked as "no pain" and the right end (100 mm) marked "worst possible pain."
Change from Baseline in ACR Core Set Values Patient's Assessment of Physical Function Using Health Assessment Questionnaire - Disability Index (HAQ-DI) | Baseline, Week 12
  Participants assess their degree of difficulty of physical function over the past week on a 4-item ordinal scale ranging from 0, "without any difficulty," to 3, "unable to do."

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- United States (20):
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Avondale, Avondale, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Flagstaff, Flagstaff, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Mesa, Mesa, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Phoenix PV, Phoenix, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Sun City, Sun City, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Tucson Southeast, Tucson, Arizona
  - Medvin Clinical Research - Covina, Covina, California
  - Newport Huntington Medical Group, Huntington Beach, California
  - Medvin Clinical Research - Tujunga, Tujunga, California
  - Medvin Clinical Research - Whittier, Whittier, California
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Willow Rheumatology and Wellness PLLC, Willowbrook, Illinois
  - Accurate Clinical Research, Inc, Lake Charles, Louisiana
  - Saint Paul Rheumatology, Eagan, Minnesota
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Accurate Clinical Management, LLC, Baytown, Texas
  - Accurate Clinical Research, Inc, Houston, Texas
  - DM Clinical Research - TRA, Tomball, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/580075